CLINICAL TRIAL: NCT01280864
Title: Investigation of Pelvic Floor-Brain Neurobiologic Axis in IC/IBS and IBS
Brief Title: MAPP Investigation of Pelvic Floor-Brain Neurobiologic Axis in IC/IBS and IBS
Status: Terminated | Type: Observational
Why Stopped: the study PI left the university of iowa
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Satish Rao, Professor, Augusta University
Other Study IDs: 200806750
Record Dates: First submitted 2011-01-19; First posted 2011-01-21 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Interstitial Cystitis; Irritable Bowel Syndrome
MeSH Terms: conditions — Cystitis, Interstitial; Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Interstitial Cystitis Alone
- Irritable Bowel Syndrome Alone
- Healthy Controls

SUMMARY:
Hypotheses:

1. The bidirectional signaling between the cortex, and the pelvic floor/gut is deranged in patients with IC and in IBS. Consequently, they will demonstrate hyperexcitability of the pelvic floor/brain axis as evidenced by shorter latencies and increased amplitudes for both the afferent anorectal-cortical evoked potentials and efferent cortically-induced (magnetic) anorectal motor evoked potentials.
2. Unlike patients with IC alone, patients with IBS will also demonstrate anorectal visceral hypersensitivity and anorectal sensory-motor dysfunction.

ELIGIBILITY:
Inclusion Criteria:Irritable Bowel Syndrome (IBS) Study Population

Inclusion criteria:

1. During the previous year, all patients must have recurrent abdominal discomfort or pain for at least 3 days per month in the last 3 months associated with two or more of the following symptoms (6): i) improvement with defecation; ii) onset associated with a change in frequency of stool; and/or iii) onset associated with a change in form (appearance) of stool (83);
2. No evidence for structural diseases (excluded by colonoscopy/ barium enema and metabolic problem by lab tests; and
3. On a prospective symptom/stool diary [Appendix 1] patients reported i) presence of abdominal pain/discomfort for at least 2 days per week; ii) hard or lumpy stools >25% and loose or watery stools in < 25% of bowel movements (IBS-C); (iii) loose or watery stools in >25% of bowel movements and hard stools <25% of BMs(IBS-D); >25% of hard or loose stools within one week (IBS-M) (6).

Exclusion Criteria:

1. Patients with laxative abuse, anorexia nervosa, and bulimia;
2. Patients taking constipating drugs, (e.g. opioids), tricyclics (because of increased seizure risk), serotonin modulators (tegaserod), antispasmodics (dicyclomine or hyoscyamine), muscle relaxants (e.g. cyclobenzaprine) unless the drug is stopped at least 2 weeks before enrollment;
3. Patients with a current history of depression and/or taking antidepressants;
4. Patients with comorbid illnesses, severe cardiac disease, chronic renal failure or previous gastrointestinal surgery except cholecystectomy and appendectomy;
5. Patients with neurologic diseases (e.g. head injuries, epilepsy, multiple sclerosis, strokes, spinal cord injuries) or brain disorders prone to causing seizures;
6. Patients experiencing impaired cognizance (mini mental score of < 15) and/or legally blind;
7. Women who are pregnant or likely to conceive (women with potential for pregnancy must use contraceptive measures to be included);
8. Patients with ulcerative and Crohns colitis;
9. Patients with rectal prolapse, anal fissure, anal surgery or inflamed hemorrhoids.

Interstitial Cystitis/Painful Bladder Syndrome (IC/PBS) Study Population

Inclusion Criteria:

IC/PBS patients who have met all three of the modified NIDDK criteria (84) for IC/PBS as described below on a urinary symptom assessment form (Appendix 3):

1. Participants will report the occurrence of bladder pain with a score of >3 on a Likert scale of 1-10.
2. Participants will report the presence of increased urinary frequency with a score of >3 on a Likert scale of 1 -10.
3. The bladder pain and increased urinary frequency will have been present for at least 6 weeks.

We recognize that the NIDDK is currently working on recommending new diagnostic criteria for interstitial cystitis. We will adopt any revised criteria commiserate with the new recommendations of the NIDDK as our study progresses.

Exclusion Criteria:

1. History of genitourinary tuberculosis, bladder cancer, high grade dysplasia, carcinoma in situ, urethra, vaginal, or cervical cancer.
2. Previous treatment with cytoxan or cyclophosphamide (as reported by the patient).
3. Radiation cystitis (as reported by the patient).
4. Neurogenic bladder dysfunction (e.g.,) due to spinal cord injury, stroke, Parkinson's, MS, spina bifida, or diabetic cystopathy (reported by the patient or determined during a neurologic exam.
5. Having had an augmentation cystoplasty (as reported by the patient).
6. Having undergone a cystectomy, cystolysis, or neuroectomy as reported by the patient.
7. Having a urethral stricture of less than 12 French (as reported by the patient).
8. Urinalysis with >10 white blood cells per high-powered field.
9. A positive urine culture for bacterial cystitis within the past three months (by report) or a positive dipstick for leucocyte esterase or nitrates on urinary dipstick test at the time of presentation.
10. Symptoms of vaginitis (as reported by the patient).
11. Active herpes at presentation or has had active herpes in the last three months (by report).
12. Use of antimicrobials in the past three months for urinary tract infections (by report).
13. Presence of bladder, ureteral, or urethral calculi (as reported by the patient).
14. Having undergone a cystometrogram, bladder cystoscopy under anesthesia or bladder biopsy under anesthesia or urethral dilation within the 6 weeks.
15. Pregnancy.

Additional Criteria for recruitment:

Patients will be assessed no sooner than 6 weeks following a DMSO or other treatment or a hydrodistention as these treatments may influence inflammation. Subjects should have had no infectious illness within 2 weeks of participation. As estrogen levels are thought to contribute to IC symptoms, and symptom exacerbation has been reported perimenstrually (85), all menstruating subjects will be tested during the mid-luteal portions of their menstrual cycle (approx. days 7-14) to control for hormonal variability.

We weighed the issue of excluding IC patients taking pain and psychotropic medication vs. including these patients. Amitriptyline is commonly used for treatment of pain in both IC and IBS; these patients commonly take other psychotropic drugs, systemic antihistamines, and drugs for pain. If we were to exclude all patients on any medication, we would be able to recruit a small and unrepresentative sample of the healthiest IC patients. If we asked patients to refrain from using medication for 2 weeks before the study, we would be subjecting them to undue pain and hardship, and might trigger an exacerbation of the disease. However, use of antihistamines affect measurements of methylhistamine, and use of amitriptyline and other anti- depressants produce a general blunting of the HPA response to a stressful stimuli (86, 87) as well as modulate the neurobiologic responses. We will exclude all subjects on antidepressants to examine a more homogeneous population. To try to obtain as representative a sample as possible without confounding of results we used the following strategy in our pilot studies and plan to use the same strategy in the proposed study. Subjects taking systemic antihistamines could not be included if they had taken antihistamines within a week of the study. Our preliminary data indicated that there was no significant difference in the ACTH or cortisol response to the reactivity challenge among patients using vs. those not using amitriptyline or other psychotropic medications (p's = .45 to .90).

Healthy Controls study population:

Additionally, we will recruit 30 healthy controls matched for our patient group with regards to age, gender, hormonal status and parity. Controls will be healthy women with no history of urological disease or genito-urinary symptoms and no immunomodulatory disease such as rheumatoid arthritis, lupus, MS, chronic fatigue, fibromyalgia, diabetes, cancer, HIV, vestibulitis, allergies, chronic fungal infections, migraines, depression, or chronic pain conditions. Healthy controls will be asked to complete the Mayo Health Screening survey and this will be used to adjudicate their health status.

Healthy controls will be on NO meds other than multivitamins, oral contraceptives, and possibly low dose aspirin. They can not be taking anti-hypertensives, serotonin reuptake inhibitors, thyroid meds or other medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects: Sixty six consecutive adult, out-patients, over 18 years with IC alone and 66 adult patients with IBS alone and 30 healthy controls will be recruited for this 5 year study and to fulfill all 4 aims of this study. All study aims will recruit under a unified strategy. For most of the funding cycle, we will recruit simultaneously for several study aims. To prevent confusion about concordant studies, similar standardized forms and diagnostic tests will be used for each aim, with supplemental tools as needed.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2010-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States